CLINICAL TRIAL: NCT03884348
Title: Helicobacter Pylori Eradication According to Sequencing-based 23S Ribosomal RNA Point Mutation Associated With Clarithromycin Resistance
Brief Title: Tailored H. Pylori Eradication Based on Clarithromycin Resistance
Status: Completed | Type: Observational
Sponsor: Kangdong Sacred Heart Hospital (Other)
Responsible Party: Principal Investigator, Shin, Woon Geon, Principal Investigator, Kangdong Sacred Heart Hospital
Other Study IDs: Kangdong2017-03-005
Record Dates: First submitted 2019-03-14; First posted 2019-03-21 (Actual); Last update posted 2019-03-21 (Actual); Status verified 2019-03

CONDITIONS: Helicobacter Pylori Infection; Antibiotic Resistant Strain
MeSH Terms: interventions — Proton Pump Inhibitors; Amoxicillin; Clarithromycin; Metronidazole

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PAM-treated clarithromycin-resistance group: Treatment with PPI twice a day, amoxicillin (1000 mg) twice a day, and metronidazole (500 mg) three times a day for 7 days in patients with clinically significant point mutations
  Interventions: Drug: proton pump inhibitor, amoxicillin, metronidazole
- PAC-treated nonresistance group: Treatment with PPI twice a day, amoxicillin (1000 mg) twice a day, and clarithromycin (500 mg) twice a day for 7 day in patients with clinically insignificant point mutations
  Interventions: Drug: proton pump inhibitor, amoxicillin, clarithromycin

INTERVENTIONS:
Drug: proton pump inhibitor, amoxicillin, clarithromycin — non-resistant group with treatment of proton pump inhibitor, amoxicillin, clarithromycin
  Groups: PAC-treated nonresistance group
Drug: proton pump inhibitor, amoxicillin, metronidazole — clarithromycin-resistant group with treatment of proton pump inhibitor, amoxicillin, metronidazole
  Groups: PAM-treated clarithromycin-resistance group

SUMMARY:
The investigators investigated the point mutations in the 23S rRNA genes of patients infected with clarithromycin-resistant H. pylori and compared the H. pylori eradication rates based on the identified clinically significant point mutations.

DETAILED DESCRIPTION:
Sequencing-based detection of point mutations identified four mutations that were considered clinically significant (A2142G, A2142C, A2143G, A2143C), while all the other mutations were considered clinically insignificant.

Participants who did not have point mutations related to clarithromycin resistance and/or had clinically insignificant point mutations were treated with PAC (proton pump inhibitor, amoxicillin, clarithromycin) for 7 days, while participants with clinically significant point mutations were treated with PAM (proton pump inhibitor, amoxicillin, metronidazole) for 7 days. H. pylori eradication rates were compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Helicobacter pylori infection

Exclusion Criteria:

* H. pylori eradication therapy within 1 year,
* antibiotics within 4 weeks,
* surgery for gastric cancer
* malignant tumors other than gastric cancer
* end-stage renal disease
* liver cirrhosis,
* pregnancy

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Helicobacter-pylori positive patients with gastritis, ulcer, adenoma
Sampling Method: Non-Probability Sample
Enrollment: 431 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Helicobacter pylori eradication rate | 2 year
  Number of participant with successful Helicobacter pylori eradication

CONTACTS AND LOCATIONS:
Overall Officials: Woon Geon Shin, Principal Investigator — Kangdong Sacred Heart Hospital

IPD SHARING:
Plan to Share IPD: No